CLINICAL TRIAL: NCT01267370
Title: Soy Polysaccharide Fiber for the Treatment of Chronic Constipation in Children: a Randomized, Double-blind Trial
Acronym: SOYFIBER
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Collaborators: Maria Eugênia Farias Almeida Motta (Unknown); Soraia Tahan (Unknown); Mauro Batista de Morais (Unknown)
Responsible Party: Mauro Batista de Morais, Universidade Federal de São Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FiberCCF-EPM1
Record Dates: First submitted 2010-12-27; First posted 2010-12-28 (Estimated); Last update posted 2010-12-28 (Estimated); Status verified 2003-10

CONDITIONS: Constipation
Keywords: clinical trial; dietary fiber; constipation; children
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Soy polysaccharide fiber (Active Comparator): Dietary fiber for treatment of chronic constipation in children
  Interventions: Dietary Supplement: Soy polysaccharide fiber
- purified soy extract, with no fiber) (Placebo Comparator): blinded control group
  Interventions: Dietary Supplement: Soy polysaccharide fiber

INTERVENTIONS:
Dietary Supplement: Soy polysaccharide fiber — Dietary Supplement: Soy polysaccharide fiber First, disimpaction was carried out with phosphate enemas for 1 to 3 days. After the children have been "cleaned out", they received a soy polysaccharide fiber supplement (powder containing 70 g of fiber/100 g) or placebo (purified soy extract, with no fiber) for 6 weeks. Fiber and placebo were given as a standard dose for the different age groups (median of 0,57 g/kg/day) - 2 to 5 years, 10 g/day; 6 to 9 years, 15 g/day; and > 10 years, 20 g/day.
  The child that had fecal impaction (a dilated rectum filled with a large amount of stool on rectal examination) during the follow-up was treated by administering phosphate enemas for 1 to 3 consecutive days.
  Arms: Soy polysaccharide fiber, purified soy extract, with no fiber
  Other Names:
  Soy polysaccharide fiber (Pró-fibra®) Purified soy extract, with no fiber (Soyac®)
  Other Names: Soy polysaccharide fiber (Pró-fibra®); Purified soy extract, with no fiber (Soyac®)

SUMMARY:
The study tested the hypothesis that soy polysaccharide fiber reduces clinical symptoms of chronic constipation.

DETAILED DESCRIPTION:
The study was performed out at outpatient clinic of Pediatric Gastroenterology at the Federal University of São Paulo (São Paulo, Brazil), located in the southeastern region of Brazil. It is a public referral hospital for pediatric gastroenterology attendance in the Metropolitan area of the São Paulo and in Brazil. In general, the patients go to consultation after a referral from a primary care center.

Study design and sample size The design was a randomized double-blind trial, placebo-controlled study. Sample size was calculated by the formula of comparison of two proportions, using clinical improvement as a primary outcome. It had been previously calculated that a minimum of 14 patients in each group will give a power of 80% to detect a effect size of 50% with significance at the level of 5% (one-sided).

ELIGIBILITY:
Inclusion Criteria:

* Patients over two years of age at first consultation and chronic functional constipation were included. Chronic constipation was defined by the occurrence of any of the following, for at least 2 weeks, independently of stool frequency: passage of hard, scybalous, pebble-like or cylindrical cracked stools, straining or painful defecation, passage of large stools that may clog the toilet, or stool frequency less than 3 per week.

Exclusion Criteria:

* The exclusion criteria applied were organic constipation, regular use of dietary fiber in the preceding 30 days or drugs causing constipation.

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2002-01; Primary Completion 2002-12 (Actual); Study Completion 2003-10 (Actual)

PRIMARY OUTCOMES:
Clinical response | 6 weeks
  Frequency of stool passage, paiful defecation, stool consistency

SECONDARY OUTCOMES:
total and segmental colonic transit time and fecal weight and moisture | 6 weeks
  Colonic transit time was evaluated by the technique of Metcalf et al. In brief, a plain abdominal radiograph performed after 24 hours from the last ingestion of 3 sets of 20 distinctive radio-opaque markers taken on 3 consecutive days. In the presence of > 20% of the markers, a further radiography was taken on the 7th day. The colonic segments were delimitated according to Arhan et al. The patients were instructed to collect the 3-day stools separately from the urine. The collected stools were used to determine the fecal weight and moisture.

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Pediatric Gastroenterology UNIFESP, São Paulo, São Paulo, Brazil